CLINICAL TRIAL: NCT01033240
Title: Clinical Study Protocol Phase 2, Randomized Study of CS-1008 in Combination With Sorafenib Compared to Sorafenib Alone as First-Line Systemic Therapy in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: CS1008- in Combination With Sorafenib Compared to Sorafenib Alone in Subjects With Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1008-A-U204
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Advanced Hepatocellular Carcinoma; Liver Cancer; Hepatic Cancer; Liver Neoplasms
Keywords: Sorafenib; CS-1008; Advanced Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — tigatuzumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Safety Cohort 1 CS-1008 and Sorafenib (Experimental): Combination of CS-1008 and sorafenib; CS-1008 (2 mg/kg per week) in combination with sorafenib (400 mg self-administered by mouth twice daily) over 4 weeks observation, and may continue treatment until progression.
  Interventions: Drug: CS-1008 2 mg/kg; Drug: Sorafenib
- Safety Cohort 2 CS-1008 and Sorafenib (Experimental): Combination of CS-1008 and sorafenib; CS-1008 (4 mg/kg per week) in combination with sorafenib (400 mg self-administered by mouth twice daily) over 4 weeks observation, and may continue treatment until progression.
  Interventions: Drug: Sorafenib; Drug: CS-1008 4 mg/kg
- Safety Cohort 3 CS-1008 and Sorafenib (Active Comparator): Combination of CS-1008 and sorafenib; CS-1008 (6 mg/kg per week) in combination with sorafenib (400 mg self-administered by mouth twice daily) over 4 weeks observation, and may continue treatment until progression.
  Interventions: Drug: Sorafenib; Drug: CS-1008 6 mg/kg
- Treatment Group 1 CS-1008 and Sorafenib (Experimental): Combination of CS-1008 and sorafenib. Treatment Group 1: CS-1008 (6 mg/kg [or as determined] loading, 2 mg/kg/week maintenance) + sorafenib twice daily (N=50)
  Interventions: Drug: Sorafenib; Drug: CS-1008 6/2 mg/kg
- Treatment Group 2 with CS-1008 and Sorafenib (Experimental): Combination of CS-1008 and sorafenib. Treatment Group 2: CS-1008 (6 mg/kg [or as determined] loading, 6 mg/kg/week [or maximum tolerated dose {MTD}] maintenance) + sorafenib twice daily (N=50)
  Interventions: Drug: Sorafenib; Drug: CS-1008 6/6 mg/kg
- Treatment Group 3 with Sorafenib Alone (Experimental): Sorafenib. Treatment Group 3: sorafenib twice daily (N=50)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: CS-1008 2 mg/kg — On a once a week basis CS-1008 will be administered intravenously starting at 2 mg/kg.
  Arms: Safety Cohort 1 CS-1008 and Sorafenib
Drug: Sorafenib — On a daily basis, one sorafenib tablet, 400 mg, is taken orally twice a day. The total daily dose of sorafenib is 800 mg. The sorafenib tablets are taken at least 1 hour before or 2 hours after a meal.
  Other Names: Nexavar
Drug: CS-1008 6/2 mg/kg — A 6 mg/kg loading dose of CS-1008 will be administered intravenously, followed by a 2 mg/kg/week maintenance dose on a once-a-week basis.
  Arms: Treatment Group 1 CS-1008 and Sorafenib
Drug: CS-1008 6/6 mg/kg — A 6 mg/kg loading dose of CS-1008 will be administered intravenously, followed by a 6 mg/kg/week maintenance dose on a once-a-week basis.
  Arms: Treatment Group 2 with CS-1008 and Sorafenib
Drug: CS-1008 4 mg/kg — On a once a week basis CS-1008 will be administered intravenously at 4 mg/kg if tolerated.
  Arms: Safety Cohort 2 CS-1008 and Sorafenib
Drug: CS-1008 6 mg/kg — On a once a week basis CS-1008 will be administered intravenously at 6 mg/kg if tolerated.
  Arms: Safety Cohort 3 CS-1008 and Sorafenib

SUMMARY:
The purpose of this study is to determine the safety and efficacy of CS-1008 in combination with sorafenib to sorafenib alone for treating liver cancer. Approximately 160 participants will take part in this study at approximately 22 sites (4 in the US, 8 in Japan, and 10 in Asia).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC) or clinical diagnosis of HCC when the following criteria are all met:

  * History of chronic hepatitis and/or cirrhosis of liver;
  * Typical features of HCC demonstrated in dynamic imaging studies, such as three-phase computed tomography (CT); AND
  * Alpha-fetoprotein (AFP) level > 200 ng/mL
* Advanced diseases

  * Extrahepatic metastasis, OR
  * Locally advanced diseases which are not amenable for surgical resection or other loco-regional therapies including transhepatic arterial (chemo) embolization (TACE or TAE) and local ablative therapy
* Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 of at least 1 untreated target lesion that can be measured in 1 dimension
* At least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Child-Pugh class A
* Life expectancy of at least 12 weeks
* Adequate organ and bone marrow function as assessed by clinical laboratory evaluations:

  * Hemoglobin ≥ 8.5 g/dL (transfusion and/or growth factor support allowed)
  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
  * Platelet count ≥ 75 x 10^9/L
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance > 40 mL/min
  * Aspartate Aminotransferase (AST) and alkaline phosphatase ≤ 5.0 x ULN
  * Total bilirubin ≤ 1.5 x ULN
* Serum amylase and lipase ≤ 1.5 x ULN
* Women of childbearing potential must be willing to consent to using effective contraception (eg, abstinence, hormonal contraceptives, bilateral tubal ligation, barrier with spermicide, intrauterine device) while on treatment and for 3 months thereafter. Men who are the partner of a woman of childbearing potential must be willing to consent to using effective contraception (eg, vasectomy or barrier with spermicide) while on treatment and for 3 months thereafter
* All female participants of childbearing potential must have a negative pregnancy test (serum or urine) result
* Participants must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an International Review Board (IRB)/ Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) before the performance of any study specific procedures or tests
* Participants must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Any prior systemic therapy for HCC, including systemic chemotherapy (prior exposure to chemotherapy by TACE is allowed), immunotherapy, sorafenib or other Raf kinase inhibitors, Vascular Endothelial Growth Factor (VEGF)/Vascular Endothelial Growth Factor Receptor (VEGFR)-inhibitors, epidermal growth factor receptor inhibitors or mechanistic target of rapamycin (mTOR) inhibitors
* Radiotherapy or major surgical procedure within 4 weeks of the screening/baseline visit or minor surgical procedures (eg, core biopsy or fine needle aspiration) within 2 weeks of the screening/baseline visit
* Anticipation of need for radiotherapy (RT) or a major surgical procedure during the study
* Any investigational agent within 4 weeks before the screening/baseline visit
* History of any of the following conditions within 6 months before the screening/baseline visit:

  * Myocardial infarction with significant impairment of cardiac function (eg, ejection fraction ≤ 30%)
  * Severe/unstable angina pectoris
  * New York Heart Association (NYHA) class III or intravenous (IV) congestive heart failure
  * Clinically significant pulmonary disease (eg, severe chronic obstructive pulmonary disease or asthma)
* Clinically active brain metastases (defined as untreated, symptomatic or requiring steroids or anticonvulsants medications to control associated symptoms), uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis. Participants with treated brain metastasis will be included in the study if they have recovered from the acute, toxic effects of radiotherapy. A minimum of 15 days must have elapsed between the end of RT and the screening/baseline visit
* History of organ transplantation
* Clinically significant, severe, active infection requiring IV antibiotics
* Known history of human immunodeficiency virus (HIV) infection
* History of prior sensitivity reaction to any components of CS-1008 or sorafenib formulations
* History of a second malignancy, with the exception of in situ cervical cancer or adequately treated basal cell or squamous cell carcinoma of the skin
* Pregnant or breast feeding
* Serious intercurrent medical illnesses that, in the opinion of the Investigator, would impair the participant's ability to provide informed consent or unacceptably reduce the safety of the proposed treatment
* Clinically significant (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] grade ≥ 3) gastrointestinal bleeding in the past 12 months or current active gastrointestinal bleeding
* Presence of esophageal varices at risk of bleeding, such as large esophageal/gastric varices or those with red sign, or active peptic ulcer with or without exposed vessels at risk of bleeding (as documented by endoscopy)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2012-07-13 (Actual); Study Completion 2013-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (28):
- United States (4):
  - Kenmar Research Group, Los Angeles, California
  - Georgetown-Lombardi Cancer Center, Washington D.C., District of Columbia
  - The Mount Sinai Medical Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Japan (9):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Hiroshima University, Hiroshima, Hiroshima
  - Kanazawa University, Kanazawa, Ishikawa-ken
  - Kinki University Hospital, Osaka, Osaka-sayama
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba University Hospital, Chiba
  - Okayama University Hospital, Okayama
  - Osaka Med Center Cancer and Cardiovascular Disease, Osaka
  - Musashino Red-Cross Hospital, Tokyo
- South Korea (7):
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Catholic Univ. of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (8):
  - Kaohiung Chang Gung Hospital, Kaohsiung City, Niaosung Hsiang
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Chiayi City
  - Kaohslung Medical University Hospital, Kaohsiung City
  - National Cheng-Kung University Hospital, Tainan
  - Chi-Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkuo, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng AL, Kang YK, He AR, Lim HY, Ryoo BY, Hung CH, Sheen IS, Izumi N, Austin T, Wang Q, Greenberg J, Shiratori S, Beckman RA, Kudo M; Investigators' Study Group. Safety and efficacy of tigatuzumab plus sorafenib as first-line therapy in subjects with advanced hepatocellular carcinoma: A phase 2 randomized study. J Hepatol. 2015 Oct;63(4):896-904. doi: 10.1016/j.jhep.2015.06.001. Epub 2015 Jun 10. PMID 26071796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 172 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at clinic sites in the United States of America (USA), Japan, Taiwan, and South Korea. Ten (10) of the participants were enrolled but did not receive treatment. The data on the 162 treated participants are presented in this report.
Groups:
- Sorafenib: Participants with advanced hepatocellular carcinoma who were administered sorafenib (400 mg) orally twice daily over 3-week treatment cycles.
- CS-1008 6/2 mg/kg + Sorafenib: Participants with advanced hepatocellular carcinoma who were administered a combination of CS-1008 (6 mg/kg loading dose followed by 2 mg/kg/week maintenance dose) intravenously (IV) once a week + sorafenib (400 mg) orally twice daily over 3-week treatment cycles.
- CS-1008 6/6 mg/kg + Sorafenib: Participants with advanced hepatocellular carcinoma who were administered a combination of CS-1008 (6 mg/kg loading dose followed by 6 mg/kg/week maintenance dose) intravenously (IV) once a week + sorafenib (400 mg) orally twice daily over 3-week treatment cycles.
Period: Overall Study
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib
Started | 55 | 53 | 55
Completed | 6 | 3 | 2
Not Completed | 49 | 50 | 53
Not completed — Serious Adverse Event (SAE) or Adverse Event | 10 | 8 | 6
Not completed — Death | 2 | 0 | 0
Not completed — Withdrew Consent | 2 | 9 | 2
Not completed — Disease Progression | 35 | 32 | 41
Not completed — Investigator Discretion | 0 | 0 | 2
Not completed — Other | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set was used to assess baseline characteristics. The full analysis set included 162 participants who were randomized and received at least one dose of sorafenib or CS-1008 in the randomized phase. All 9 participants in the safety cohort portion of the study were discontinued after the primary analysis cut-off date and not included in the randomized portion with the full analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib | Total
Number analyzed (Participants) | 55 | 53 | 54 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (11.36) | 60.7 (12.92) | 61.1 (12.47) | 62.4 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 28
  Male | 44 | 45 | 45 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 32 | 37 | 103
  Unknown or Not Reported | 21 | 21 | 17 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 54 | 52 | 53 | 159
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 0 | 1 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 20 | 15 | 18 | 53
  United States | 1 | 1 | 1 | 3
  Japan | 17 | 17 | 18 | 52
  Taiwan | 17 | 20 | 17 | 54

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) Following CS1008 in Combination With Sorafenib Compared to Sorafenib Alone in Participants With Advanced Liver Cancer
Description: Time to progression was defined as the time from randomization to the date of the first objective documentation of radiographic or symptomatic progression, whichever came first.
Time Frame: Baseline up to approximately 2 years post-dose.
Population: The full analysis set was used to assess TTP.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib
Number analyzed (Participants) | 55 | 53 | 54
months | 2.8 [1.5 to 6.6] | 3.0 [2.6 to 5.5] | 3.9 [2.7 to 5.3]

2. Secondary Outcome: Overall Survival Following CS1008 in Combination With Sorafenib Compared to Sorafenib Alone in Participants With Advanced Liver Cancer
Description: Overall survival (OS) was defined as the time from randomization to the date of death. The factors in the final model were treatment, Eastern Cooperative Oncology Group (ECOG) performance status, presence of extrahepatic metastasis and/or macrovessel invasion, and region.
Time Frame: Baseline up to approximately 3 years 2 months post-dose.
Population: The full analysis set was used to assess overall survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib
Number analyzed (Participants) | 55 | 53 | 54
months | 8.2 [4.9 to 13.4] | 8.2 [5.7 to 10.4] | 12.2 [9.0 to 15.0]

3. Secondary Outcome: Best Overall Response and Objective Response Rate Following CS1008 in Combination With Sorafenib Compared to Sorafenib Alone in Participants With Advanced Liver Cancer
Description: The best overall response is the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], unconfirmed CR, unconfirmed PR, stable disease [SD], and progressive disease [PD]) among all overall responses recorded from the start of treatment until the participant withdraws from the study based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. If there is no tumor assessment after the first dose of study drug, the best overall response is classified as Inevaluable. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD defined as at least a 20% increase in the sum of diameters of target lesions. Objective response rate was defined as confirmed CR and confirmed PR.
Time Frame: Baseline up to disease progression, death, lost to follow up, or study discontinuation (whichever comes first), up to approximately 3 years 2 months post-dose.
Population: The full analysis set was used to assess the best overall response and objective response rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib
Number analyzed (Participants) | 55 | 53 | 54
Participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 6 | 3 | 8
  Objective Response Rate (CR+PR) | 6 | 3 | 8
  Stable Disease (SD) | 24 | 26 | 29
  Progressive Disease (PD) | 20 | 14 | 15
  Inevaluable | 5 | 10 | 2
  Best Overall Response of SD or Better | 30 | 29 | 37

4. Secondary Outcome: Treatment-Emergent Adverse Events Following CS1008 in Combination With Sorafenib Compared to Sorafenib Alone in Participants With Advanced Liver Cancer
Description: Treatment-Emergent Adverse Events (TEAEs) were defined as those adverse events (AEs) that occurred, having been absent before the study, or worsened in severity after the initiation of study treatment administration. An AE that occurred more than 30 days after the last dose of study medication was not included as a TEAE unless it was considered related to treatment or the assessment of relatedness was missing.
Time Frame: Baseline up to 30 days after last dose, up to approximately 3 years 2 months post-dose.
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib
Number analyzed (Participants) | 55 | 52 | 55
Participants
  Subjects with ≥1 TEAE | 54 | 52 | 54
  TEAEs by worst CTCAE grade: CTCAE grade: Grade ≥ 3 | 43 | 44 | 46
  TEAEs by worst CTCAE grade: Grade 5 | 10 | 8 | 5
  TEAEs related to CS-1008 | NA — Twelve participants in the sorafenib-only group were mistakenly reported as having experienced TEAEs related to CS-1008. Confirmation from the sites that these participants never received CS-1008. | 40 | 39
  TEAEs related to sorafenib | 53 | 51 | 54
  Discontinued CS-1008 due to TEAE | 0 | 5 | 8
  Discontinued sorafenib due to TEAE | 18 | 7 | 9
  Treatment-Emergent SAEs | 25 | 26 | 20
  TEAEs leading to death | 11 | 8 | 6
  Deaths | 34 | 31 | 29

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) data were collected from Baseline up to 30 days after the last dose, up to approximately 3 years 2 months post-dose.
Description: Treatment-Emergent Adverse Events (TEAEs) were defined as those adverse events (AEs) that occurred, having been absent before the study, or worsened in severity after the initiation of study treatment administration. An that occurred >30 days after last dose of study medication was not included as a TEAE unless it was considered related to treatment or the assessment of relatedness was missing.
Arm/Group | Sorafenib | CS-1008 6/2 mg/kg + Sorafenib | CS-1008 6/6 mg/kg + Sorafenib
All-Cause Mortality (participants affected / at risk) | 34/55 | 31/52 | 29/55
Serious Adverse Events (participants affected / at risk) | 25/55 | 26/52 | 20/55
Other Adverse Events (participants affected / at risk) | 54/55 | 52/52 | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=55) | CS-1008 6/2 mg/kg + Sorafenib (N=52) | CS-1008 6/6 mg/kg + Sorafenib (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 6 | 6 | 5
Fatigue (General disorders) | 1 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic infarction (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0
Blood amylase increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Decreased appetitie (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 4 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=55) | CS-1008 6/2 mg/kg + Sorafenib (N=52) | CS-1008 6/6 mg/kg + Sorafenib (N=55)
Anaemia (Blood and lymphatic system disorders) | 6 | 5 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5 | 6
Tinnitus (Ear and labyrinth disorders) | 4 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 4 | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 10 | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 12 | 14 | 17
Abdominal pain upper (Gastrointestinal disorders) | 3 | 10 | 13
Ascites (Gastrointestinal disorders) | 14 | 14 | 7
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 9 | 19 | 13
Diarrhoea (Gastrointestinal disorders) | 27 | 23 | 36
Dry Mouth (Gastrointestinal disorders) | 5 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 7
Gingival bleeding (Gastrointestinal disorders) | 3 | 3 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 10 | 11
Stomatitis (Gastrointestinal disorders) | 6 | 5 | 6
Vomiting (Gastrointestinal disorders) | 7 | 5 | 10
Asthenia (General disorders) | 5 | 6 | 3
Chills (General disorders) | 3 | 5 | 4
Disease progression (General disorders) | 6 | 6 | 5
Fatigue (General disorders) | 17 | 13 | 14
Malaise (General disorders) | 6 | 6 | 7
Oedema peripheral (General disorders) | 11 | 14 | 10
Pyrexia (General disorders) | 9 | 16 | 15
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 5
Pneumonia (Infections and infestations) | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 8 | 5
Alanine aminotransferase increased (Investigations) | 14 | 14 | 15
Aspartate aminotransferase increased (Investigations) | 24 | 20 | 21
Blood alkaline phosphatase increased (Investigations) | 5 | 3 | 9
Blood amylase increased (Investigations) | 8 | 12 | 11
Blood bilirubin increased (Investigations) | 13 | 12 | 9
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 7
Blood creatinine increased (Investigations) | 4 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 6 | 5 | 7
Blood urea increased (Investigations) | 3 | 3 | 1
Lipase increased (Investigations) | 19 | 17 | 17
Lymphocyte count decreased (Investigations) | 4 | 8 | 10
Neutrophil count decreased (Investigations) | 4 | 1 | 3
Platelet count decreased (Investigations) | 14 | 8 | 15
Weight blood cell count decreased (Investigations) | 4 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 25 | 25 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 12 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 17 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 11
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 5 | 4 | 2
Dysgeusia (Nervous system disorders) | 3 | 1 | 2
Headache (Nervous system disorders) | 4 | 8 | 9
Hepatic encephalopathy (Nervous system disorders) | 4 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 5 | 8 | 11
Proteinuria (Renal and urinary disorders) | 2 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 14 | 14 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 19 | 18
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5 | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 7 | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 35 | 37 | 42
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7 | 9
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 3 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 20 | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No